CLINICAL TRIAL: NCT04598958
Title: A Multidisciplinary "Integrated Management Team to Improve Maternal-Child Outcomes (IMPROVE)" Intervention to Improve Maternal and Child Outcomes and HIV Service and Antiretroviral Therapy Uptake and Retention in Lesotho
Brief Title: A Multidisciplinary "Integrated Management Team to Improve Maternal-Child Outcomes (IMPROVE)" Intervention to Improve Maternal and Child Outcomes in Lesotho
Acronym: IMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Ministry of Health, Lesotho (Other Government); United States Agency for International Development (USAID) (U.S. Federal Agency); Avenir Health (Unknown); Population Council (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EG0142
Record Dates: First submitted 2020-10-05; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Human Immunodeficiency Virus
Keywords: maternal child health; prevention of mother to child transmission; HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized design. Two clusters of health facilities were randomized to receive either the intervention or standard of care. There are 6 facilities in each cluster. Individual participants are treated based on the cluster they fall into
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMPROVE (Experimental): A cluster of 6 health facilities are to receive the IMPROVE Intervention. The IMPROVE intervention includes: (1) Multidisciplinary integrated management teams to coordinate patient-focused and outcome-oriented PMTCT and MCH services; (2) Enhanced Positive Health, Dignity, and Prevention (PHDP)-focused counseling and skills-building training and job aids; and (3) Increased early community-based counseling and support for first (antenatal care clinic) ANC attendees with particular attention to HIV-positive women to minimize loss to follow-up.
  Interventions: Other: IMPROVE
- Standard of care (No Intervention): A cluster of 6 health facilities receive Standard of Care. Routine health facility services offering the national standard of care for pregnant and breastfeeding women in Lesotho

INTERVENTIONS:
Other: IMPROVE — Health system interventions that include: (1) Multidisciplinary integrated management teams to coordinate patient-focused and outcome-oriented PMTCT and MCH services; (2) Enhanced Positive Health, Dignity, and Prevention (PHDP)-focused counseling and skills-building training and job aids; and (3) Increased early community-based counseling and support for first (antenatal care clinic) ANC attendees
  Arms: IMPROVE

SUMMARY:
This study aims to improve maternal and child health (MCH) outcomes by implementing and evaluating a multidisciplinary "Integrated Management Team to Improve Maternal-Child Outcomes (IMPROVE)" intervention to increase MCH, antiretroviral therapy (ART), and HIV services uptake and retention in Lesotho. The proposed intervention will focus efforts to improve the effectiveness of existing village health workers (VHW) and HIV support organizations (Lesotho Network of AIDS Service Organizations [LENASO] and Mothers2Mothers [M2M]) based at the facility and coordination between the facility and community. The IMPROVE intervention includes: (1) Multidisciplinary integrated management teams to coordinate patient-focused and outcome-oriented PMTCT and MCH services; (2) Enhanced Positive Health, Dignity, and Prevention (PHDP)-focused counseling and skills-building training and job aids; and (3) Increased early community-based counseling and support for first (antenatal care clinic) ANC attendees with particular attention to HIV-positive women to minimize loss to follow-up.

The study will be a cluster randomized design with facilities randomized to receive the IMPROVE intervention or routine services offering the national standard of care. A cohort of HIV-positive and HIV-negative pregnant women will be enrolled and prospectively followed every three months through pregnancy and until the participant's child reaches 24 months of age. The primary HIV objectives will be to evaluate the effect of the intervention on retention in HIV care, viral suppression, adherence to ART in HIV-positive women, and HIV retesting in HIV-negative women. The investigators will also assess the effect of the IMPROVE intervention on general MCH indices including antenatal care (ANC) attendance, facility delivery, family planning, and immunization coverage. Secondary objectives include evaluation of adherence self-efficacy (HIV positive) or prevention self-efficacy (HIV negative), depression and stigma as well as disclosure, knowledge of partner status, and identification of discordant couples in intervention versus control facilities. Analysis of the cost-effectiveness of the IMPROVE intervention will also be conducted. In addition, qualitative interviews and focus group discussions will be conducted with study women, health care workers (HCW), LENASO, and VHWs to evaluate the feasibility and acceptability of integrating this intervention into routine care.

DETAILED DESCRIPTION:
Lesotho is among countries with the highest HIV prevalence worldwide, with an estimated prevalence of HIV among pregnant women of 25.8% in 2013. In April 2013, Lesotho transitioned from the WHO "Option A" strategy to implementation of "Option B+" (lifelong ART for all HIV-positive women) strategy for PMTCT, in the context of a program that is integrated into MCH services. Through this study, the investigators propose to evaluate a package of interventions to provide enhanced individualized counseling and community support within a coordinated system of training and accountability to optimize the delivery of patient-focused services using PHDP principles within the routine PMTCT/MCH program in Lesotho.

The study will be conducted in 12 health facilities in Maseru district.

The proposed intervention will focus efforts to improve the effectiveness of existing VHW and HIV support organizations (LENASO, M2M) based at the facility and coordination between the facility and community. The package includes:

1. MCH staff, counselors, M2M/LENASO and VHWs meeting regularly to coordinate patient-focused and outcome-oriented PMTCT and MCH services to all women, with immediate follow-up of defaulters.
2. Enhanced Positive Health, Dignity, and Prevention (PHDP)-focused counseling and skills-building training and job aids to improve the quality and consistency of counseling provided by all IMPROVE team members. Such individualized support will facilitate self-efficacy, support partner disclosure, provide screening and referral for depression, and provide linkages to community-based services.
3. Increased early community-based counseling and support for all ANC attendees that will include 1 to 2 additional home or community visits at 2-7 days and/or 9-14 days after first ANC visit, with particular attention to HIV-positive women to minimize immediate and early loss to follow-up (LTFU).

Aim and Objectives: The overall aim of this study is to improve maternal and child health outcomes by implementing and evaluating a multidisciplinary "Integrated Management Team to Improve Maternal-Child Outcomes (IMPROVE)" intervention to increase overall MCH, ART, and HIV service uptake and retention.

Primary Objectives:

1. To evaluate the effect of the IMPROVE intervention on retention in HIV care, viral suppression, and adherence to ART at 24 months postpartum in a prospective cohort of HIV-positive pregnant/postpartum women and their infants compared to a cohort of HIV-positive women receiving routine care alone.
2. To evaluate the effect of the IMPROVE intervention on repeat HIV testing by 24 months postpartum in a prospective cohort of HIV-negative pregnant/postpartum women compared to a cohort of HIV-negative women receiving routine care alone.
3. To evaluate the effect of the IMPROVE intervention on targeted MCH health seeking behaviors (e.g., facility delivery, child immunization) in both HIV-positive and HIV-negative women compared to women receiving routine care alone.
4. To determine the costs associated with the IMPROVE package of interventions for both HIV-positive and HIV-negative women compared to HIV-positive and HIV-negative women receiving routine care without the IMPROVE intervention.

Secondary Objectives:

1. To assess additional MCH outcomes (e.g., ANC attendance, infant mortality, maternal mortality); other HIV prevention indices (e.g., disclosure, knowledge of partner status, identification of discordant couples); unintended pregnancy prevention indices (e.g., use of modern contraceptives, repeat pregnancy, fertility intentions); and other indices of HIV care (e.g., timing of infant diagnosis, number of infected infants) among HIV-positive and HIV-negative women receiving the IMPROVE intervention versus those receiving routine care alone.
2. To compare depression, experienced stigma, and self-efficacy among both HIV-positive (treatment self-efficacy) and HIV-negative women (HIV prevention self-efficacy) in the intervention and control facilities.
3. To compare pregnant/postpartum women's attitudes toward lifelong ART (HIV-positive only), acceptability of the IMPROVE intervention (intervention facilities only), and satisfaction with PMTCT/MCH services among both HIV-positive and HIV-negative women in intervention and control facilities.
4. To assess HCW, counselor, and VHW attitudes toward the feasibility and acceptability of integrating the IMPROVE package in routine services.
5. To evaluate the cost-effectiveness of the IMPROVE intervention on retention in HIV care, viral suppression and adherence to ART, HIV retesting, and uptake of family planning and child immunizations at 24 months postpartum in a prospective cohort of pregnant/postpartum women and their infants compared to a similar cohort of women and infants receiving routine care without the IMPROVE intervention.

Hypotheses:

1. HIV-positive women in facilities with IMPROVE versus routine care will have higher adherence and retention in HIV care.
2. HIV-negative women in facilities receiving the IMPROVE intervention will have an increase in HIV re-testing in the postpartum period.
3. HIV-positive and HIV-negative women in facilities with IMPROVE versus routine care will show improvement in health seeking behavior, leading to improved maternal and infant outcomes.
4. The IMPROVE intervention is a cost-effective approach to improve health outcomes among HIV-positive and HIV -negative pregnant/postpartum women and their infants.

Data gathering activities: The study will be conducted in Maseru district, which is large and representative of a variety of settings within Lesotho. Maseru has one of the highest HIV prevalence rates and the lowest PMTCT and MCH indicator coverage rates in Lesotho. Twelve health facilities serving between 150-900 pregnant women annually from Maseru district were purposefully selected to reflect a common range of ANC volumes while allowing for timely recruitment of the sample size of HIV-positive women needed during the enrollment period. Pregnant women attending their first ANC visit at a study health facility will be eligible for enrollment in a prospective cohort and followed until 24 months' post-partum. Because the study intervention begins at the first ANC visit with enhanced counseling and close follow-up at home within the next week, the study will only enroll women who are attending ANC for their first visit. The investigators will enroll ~310 HIV-positive and 200 HIV-negative women in each arm over 10-15 months, for a total of 1020 participants.

After obtaining written informed consent, pregnant women will be enrolled in the study into either the IMPROVE intervention arm or control arm depending on the facility the woman attends. At enrollment, women will undergo an interview to collect demographic, pregnancy, medical and HIV related information. Clinical and laboratory data will be abstracted from clinic medical records. After the enrollment visit, women/infants will be seen by study staff for study specific visits during ANC at the next ANC visit after enrollment or sooner if late in gestation (timing depends on gestational age at first visit), around the time of delivery, 6 and 14 weeks and 6, 9, 12, 18, and 24 months postpartum. Study visits will be scheduled to coincide with routine health service visits to the clinic for the mother or child as much as possible. At each study visit, a participant interview and abstraction of clinical and laboratory data from medical records will be conducted.

Study nurses will be present in each study facility and will be responsible for the collection and maintenance of study records and data. Informed consent documents, study screening/enrollment logs, and participant locator forms that include identifiable information will be completed at enrollment and stored in a locked secure location in the health facility with access limited to study staff. Multivariate random-effects 2-stage model (level-1: individual, level-2: cluster) logistic regression will be used to compare proportional outcomes between intervention and control groups. Time to event outcomes will be analyzed using survival analysis approaches. An "intent to treat" analysis will be used. Descriptive analyses will be used for the assessment of the fidelity to the IMPROVE intervention implementation over time and secondary outcomes that are likely to be infrequent and thus with limited power to detect differences (such as mortality, HIV infection rates in children, seroincidence, repeat pregnancies, etc.) The evaluation results will be presented as either odds ratios or hazard ratios (for the time-to-event analysis), and 95% confidence intervals.

Risks and Benefits to Participants: There may or may not be direct benefits to study participants. However, possible benefits to the participants include close monitoring that may identify problems sooner, screening and referral for depression, additional viral load monitoring for HIV-positive women, and potential receipt of improved service delivery for women in IMPROVE intervention facilities.

The study poses minimal safety risks to the study participants. The services are being conducted in the framework of routine MCH services. The intervention addresses mainly service delivery changes that do not subject study participants to risks outside of what would be expected within routine services. Potential risks include the potential for unintended disclosure of mother and infant's HIV status. All efforts will be made to conduct interviews in private to protect participant confidentiality.

Women enrolled in the IMPROVE study will be identified by their unique study identifier, and data collection and forms will be linked to the patient using this unique identifier only. Study participants will not receive any compensation or incentive for participating in the study.

Qualitative data collection: A subset of women participating in the study (~ 40 in each arm) will be asked to undergo semi-structured interviews for a total of about 80 semi-structured interviews. These will include approximately 20 HIV-positive and 20-HIV negative women in each of the intervention and control arms. Women attending their 18 or 24 month visit during the time that the qualitative component is underway will be randomly selected to participate in a semi-structured interview. Focus Group Discussions (FGDs) will be used to gather information about the HCW and VHW/LENASO/M2M experiences, with separate FGD for the two cadres. Sources of qualitative data will be the open-ended responses from interviews and FGDs. All qualitative data will be entered into Microsoft Word as data files and analyzed using MAXqda or another similar qualitative data analysis program. Prior to beginning study procedures for this component of the study, verbal informed consent will be documented for all individuals participating in interviews by study staff trained in protocol and ethical procedures.

Costing data collection: The cost-effectiveness component of the study will measure the cost-effectiveness of the IMPROVE intervention in achieving positive health outcomes among pregnant/postpartum women and their infants. The endpoints of the study relevant to the cost-effectiveness analysis are: 1) retention through 24 months postpartum 2) ART adherence among HIV-positive women, 3) viral load suppression among HIV-positive women 4) rate of HIV re-testing among HIV-negative women (5) rate of family planning uptake (6) rate of immunization uptake. These will be among the inputs used to compute Quality of Life Years (QALYs) gained per woman.

The outcomes will be measured in terms of incremental cost per QALY gained per HIV-positive woman, cost per infection averted per HIV-exposed infant, cost per QALY gained per HIV exposed infant, cost per adult HIV infection averted, cost per birth averted, and cost per child death averted.

The outcomes will be computed using the OneHealth Tool and data compiled from the primary endpoints. The cost estimation will include a summation of the IMPROVE intervention package plus the sum of costs incurred by participants (pregnant and postpartum women and infants) for service provision less any cost savings achieved through (1) productivity losses averted and (2) costs averted per treatment (or prevention) of disease.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman attending first ANC visit at a study facility . There is no age restriction for study enrollment as young pregnant women in Lesotho are consider emancipated.

  * HIV status known at time of enrollment
  * Residing in an area around a study facility
  * Willing and able to provide informed consent

Exclusion Criteria:

* Pregnant women attending 2nd or later ANC visits
* Attending care at study facility temporarily
* Significant medical or psychological condition that would preclude active study participation
* Inability to provide informed consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1004 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Retention | at 24 months post partum
  Proportion of participants retained in care
ART Adherence | at 24 months postpartum
  Proportion of HIV-positive women on treatment with >95% adherence based on effective pill count
Viral suppression rate | at 24 months postpartum
  Proportion of HIV-positive women with undetectable viral load
HIV retesting rate | at 24 months postpartum
  Proportion of HIV-negative women who received additional HIV testing
Targeted MCH health seeking behaviors | At 24 months postpartum
  Proportion of women who delivered at a health facility

SECONDARY OUTCOMES:
General MCH Outcomes | 24 months postpartum
  Maternal and infant survival
HIV outcomes | at 6 weeks of infant age
  Proportion of HIV exposed infants undergoing HIV testing
  Proportion of HIV exposed infants undergoing HIV testing and proportion who are HIV infected
Depression | at enrollment
  Proportion of women with depression based on Patient Health Questionnaire (PHQ-9)
Cost-effectiveness of implementing the IMPROVE intervention | At 24 months postpartum
  Incremental cost per QALY gained per HIV-positive woman and Cost per infection averted per HIV-exposed infant

CONTACTS AND LOCATIONS:
Overall Officials: Appolinaire Tiam, MD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation; Laura A Guay, MD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation; Lynne Mofenson, MD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation; Vincent Tukei, MD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation

IPD SHARING:
Plan to Share IPD: No
The dataset generated and used for this analysis is available from the study biostatistician (hhoffman@gwu.edu) on reasonable request

REFERENCES:
- [Derived] Beres LK, Chabela M, Masitha M, Catanzarite Z, Tukei VJ, Mofenson L, Tiam A, Greenberg L, Mokone M, Thabelo R, Nchephe M, Mots'oane T, Guay L, Knowlton AR. An integrated, multidisciplinary management team intervention to improve patient-centeredness, HIV, and maternal-child outcomes in Lesotho: formative research on participatory implementation strategies. BMC Health Serv Res. 2024 Dec 18;24(1):1590. doi: 10.1186/s12913-024-12049-x. PMID 39696296